CLINICAL TRIAL: NCT04498312
Title: Comparison of Extracorporeal Shock Wave Therapy Versus Manual Lymphatic Drainage on Cellulite Post Liposuction
Brief Title: Extracorporeal Shock Wave Therapy Versus Manual Lymphatic Drainageon Cellulite Post Liposuction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68mn
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite | interventions — Extracorporeal Shockwave Therapy; Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock wave group (Experimental): Received Extracorporeal shock wave therapy twice/week for 4 weeks
  Interventions: Other: Extracorporeal shock wave
- Manual lympharic group (Experimental): Received manual lymphatic drainage twice a week for four weeks
  Interventions: Other: Extracorporeal shock wave

INTERVENTIONS:
Other: Extracorporeal shock wave — The participant was placed into supine lying position then the head of the shock wave was applied on the anterior or posterior aspect of the thigh which was scanned with 2000 shots for both horizontal direction and vertical direction. The period of each session was 15 minutes, 2 times/week for 4 weeks
  Other Names: Manual lymphatic drainage

SUMMARY:
To determine whether extracorporeal shock wave therapy (ESWT) or manual lymphatic drainage (MLD) is more effective for decreasing post-liposuction cellulite.

Thirty females with grade 3 cellulite were randomly distributed into two equal groups: group A (ESWT group) (n=15) and group B (MLD group) (n=15). The cellulite grade was assessed by using the cellulite grading scale, and the thickness of subcutaneous fat was assessed by the skinfold caliper. The assessment was carried out before starting the treatment and after 4 weeks. All participants received treatment 2 times/ week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* age ranged from 25-45 years old,
* non- pregnant females
* grade 3 cellulite at thigh area after liposuction

Exclusion Criteria:

* Breastfeeding females
* Inflammatory skin disorders in the treatment area
* Edema
* Varicose veins-
* Any therapy or disease that may affect treatment

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Cellulite grade | 4 weeks
  Cellulite grading scale grade 0: means a smooth surface of the skin while standing, grade 1: means mattress phenomena upon pinch-test, grade 2: means mattress phenomena spontaneously while standing, grade 3: means mattress phenomena while in standing and lying position Higher score means bad progression

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided